CLINICAL TRIAL: NCT05124327
Title: Compliance and Satisfaction With a Remote Postpartum Vital Sign Monitoring and Follow-up Program for Hypertensive Disorders of Pregnancy (HDP) for 10 Days Postpartum
Brief Title: Remote Monitoring and Follow-up for Postpartum Hypertensive Disorders of Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Margo B. Minissian, Executive Director, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001570
Record Dates: First submitted 2021-10-01; First posted 2021-11-17 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Hypertensive Disorder of Pregnancy; Preeclampsia; Gestational Hypertension
Keywords: Remote monitoring; Hypertension; Pregnancy; HDP; RPM; Telemedicine
MeSH Terms: conditions — Toxemia; Pre-Eclampsia; Hypertension, Pregnancy-Induced; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Other): Implementation of quality improvement initiative to utilize RPM in PP HDP. Patients will utilize remote monitoring technology and bluetooth enabled BP buff to self monitor BPs- autopopulate to provider portal, and then have a telemedicine appointment at 48 hours post hospital discharge.
  Interventions: Other: QI project- usage of RPM

INTERVENTIONS:
Other: QI project- usage of RPM — close monitoring through RPM to analyze feasibility and compare readmission rates

SUMMARY:
The literature unequivocally supports follow-up in the postpartum period post hospital discharge in hypertensive patients, compared to uncomplicated delivery follow-up recommendations of 4-6 weeks postpartum, leading to decreased morbidity and mortality, utilizing at-home blood pressure monitoring and virtual/telemedicine appointments. There is much evidence that telemedicine visits are equally, if not more effective, result in cost savings, and are generally preferred by patients, specifically when there is a risk of exposure for the patient and newborn, an appropriate factor to consider amidst the global Covid-19 pandemic. Maternal health and well-being have substantial links with cultural and racial factors. Black women are three times as likely to have morbid outcomes related to gestational complications, specifically hypertensive disorders of pregnancy. Minority populations have historically displayed inferior access to care due to concerns related to transportation, healthcare insurance, or provider accessibility and distrust, resulting in diminished compliance with follow-up and negative health sequelae.

Telemedicine follow-up within 10 days of delivery (48-72 hours after discharge) reduces readmission rates, increase access to- and compliance with care, and improve patient safety satisfaction, thus establishing feasibility. Home vital sign monitoring gives an increased volume of data points for providers to utilize in titrating antihypertensive medications to optimize blood pressure control, ultimately decreasing stroke and cardiovascular risk. Existing research lacks comprehension regarding specific cardiological impacts of labile postpartum blood pressures, however researchers inferentially hypothesize that poor blood pressure management in the postpartum period can have devastating long-term cardiological consequences.

This QI project will demonstrate standardized programming for patients with hypertensive disorders of pregnancy (HDP), which may potentially lead to increased compliance, satisfaction, and accessibility, resulting in improved long-term cardiovascular health in vulnerable populations. The American heart Association (AHA) and ACOG have established that HDP are associated with long-term cardiovascular disease, however obstetricians lack guidance on effective, evidence-based research for standardization of care, leading to subsequently disjointed medical management with much room for error in transitioning from obstetrician to internist or cardiologist. Thus, implementing and establishing feasibility of remote monitoring and follow-up while applying standardized algorithms and protocols for antihypertensive medication titration and management may provide support in addressing and eradicating these gaps. As such, this pilot project has massive prospective future applicability and benefit for a highly vulnerable population.

DETAILED DESCRIPTION:
This QI project out of CSMC will create a formal remote patient follow-up and monitoring program utilizing the platform Vytrack as its' primary technology. Vytrack has the capability to sync with the EHR utilized by CSMC (C-S Link, an iteration of Epic), however this feature will not be utilized in establishing feasibility during this pilot project, due to cost prohibitions. Vytrack will provide participants with Bluetooth technology that automatically uploads in real-time and access to an application on participant's personal smartphone devices. Providers may choose to create emergency alerts within desired parameters for participant's uploaded vital signs via a provider portal.

30 participants will be manually enrolled with Vytrack after eligibility is confirmed by the primary investigator. Participants will receive standard education on how to properly use Vytrack technology and prompted to check their vital signs twice daily (morning and night) or more per primary obstetrician preference until the end of their enrollment period (ten days postpartum), while additionally maintaining their primary obstetrician's standard care. Additionally, participants will be scheduled for a virtual medical appointment at 48-72 hours post hospital discharge for vital sign evaluation and optimization with a provider, employing an algorithm to titrate antihypertensive therapy as needed. The initial usage of antihypertensive therapy will be in accordance with the participant's care team as an inpatient.

The goal of this project is predominantly to establish feasibility of such programming in this large academic hospital setting through ascertaining retention rates over ten days postpartum as well as participant satisfaction, with a target of at least 90% retention and compliance rate and at least 80% satisfaction over traditional methods. Satisfaction will be analyzed through post-participation surveys, displaying Likert-scale style questions. Secondarily, through improved patient engagement in postpartum care and accessibility to standardized management, this QI project anticipates at least a 20% reduction in postpartum readmissions for hypertensive emergencies.

ELIGIBILITY:
Inclusion Criteria:

* postpartum hypertensive women
* aged 18 years or greater
* in the hospital after delivery
* any documented concern related to blood pressure elevation including preeclampsia, gestational hypertension, essential/chronic/pregestational hypertension, or new onset postpartum hypertension
* with or without lab abnormalities
* any gestational age
* English-speaking
* access to a smartphone device

Exclusion Criteria:

* patients with eclampsia
* documented HELLP syndrome (hemolysis, elevated liver enzymes, low platelets)
* patients requiring a massive transfusion protocol (MTP)
* patients who underwent hysterectomies
* patients that were admitted to the ICU after delivery and patients who experienced fetal demise.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — postpartum patients
Enrollment: 30 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with RPM compared with standard of care | through 10 days postpartum
  Patient satisfaction with remote patient monitoring as measured by designed satisfaction surveys (not yet validated) after intervention. Survey is Likert style scale, each response is associated with a value
Adherence with the program | ten days postpartum
  volume of patients that are compliant with providing study measurements- i.e submit vital signs in VyTrac application twice a day for enrollment period

SECONDARY OUTCOMES:
Readmission rate | through 6 weeks postpartum
  postpartum readmission for hypertensive crises
Out of range blood pressures | through 10 days postpartum
  blood pressures that are outside of the normal range (above 160/110)
titration of blood pressure medication | within 10 days postpartum
  how many times antihypertensives needed to be titrated

CONTACTS AND LOCATIONS:
Overall Officials: Leah Spiro, FNP, Study Director — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ACOG — https://www.acog.org/-/media/project/acog/acogorg/clinical/files/committee-opinion/articles/2018/05/optimizing-postpartum-care.pdf
- See also: Assad, N., Drewry, A., Hoppe, K.K., Passmore, S.R., Thomas, N.A. (2021). Patient perceptions, opinions and satisfaction of telehealth with remote blood pressure monitoring postpartum. BMC Pregnancy Childbirth, 21: 153 — http://dx.doi.org/10.1186/s12884-021-03632-9
- See also: Attenello, F.J., D'Alton, M., Friedman, A.M., Goffman, D., Mack, W.J., Wen, T., & Wright, J.D. (2019). Hypertensive postpartum admissions among women without a history of hypertension or preeclampsia. Obstetrics and Gynecology, 133(4), 712-719. — http://dx.doi.org/10.1097/AOG.0000000000003099
- See also: Beigi, R.H., Binstock, A., Hauspurg, A., Hyagriv, S.N., Larkin, J., Lemon, L., Watson, A.R., & Quinn, B.A. (2019). A postpartum remote hypertension monitoring protocol implemented at the hospital level. Obstetrics & Gynecology, 134(4), 685-691. — http://dx.doi.org/10.1097/AOG.0000000000003479
- See also: Early postpartum discharge during the COVID-19 pandemic. Journal of Perinatal Medicine, 48(9), 1008-101 — http://dx.doi.org/10.1515/jpm-2020-0337
- See also: Castleman, J.S., Ganapathy, R., Grewal, A. (2016). Remote monitoring of blood pressure to reduce the risk of preeclampsia related complications with an innovative use of mobile technology. Pregnancy Hypertension, 6(4), 263-264. — http://dx.doi.org/10.1016/j.preghy.2016.04.005
- See also: Telehealth with remote blood pressure monitoring for postpartum hypertension: A prospective single-cohort feasibility study. Pregna — https://pubmed.ncbi.nlm.nih.gov/30825917/
- See also: Exploring implementation of m-health monitoring in postpartum women with hypertension. Telemedicine Journal and E-Health, 23(10), 8 — https://pubmed.ncbi.nlm.nih.gov/28475431/
- See also: Lackan, N. A., Lykens, K., Mains, D.A., Sammer, C.E., & Singh, K.P. (2010). What is patient safety culture? A review of the literature. Journal of Nursing Scholarship, 42(2), 156-165. — https://pubmed.ncbi.nlm.nih.gov/20618600/
- See also: McFarlin, B.L., Mogos, M.F., Salemi, J. L., Salihu, H.H., & Spooner, K.K. (2018). Hypertensive disorders of pregnancy and postpartum readmission in the United States national surveillance of the revolving door. Journal of Hypertension, 36(3), 608-618. — http://dx.doi.org/10.1097/HJH.0000000000001594